CLINICAL TRIAL: NCT01532934
Title: The Impact of Psychopathic Traits on the Efficacy of a Brief Intervention for Substance Use
Brief Title: The Impact of Psychopathic Traits on the Efficacy of a Substance Use Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, MarcSwogger, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28780; K23DA027720 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-15 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance Use; Psychopathy
Keywords: substance use; psychopathy; motivational enhancement; criminal recidivism
MeSH Terms: conditions — Substance-Related Disorders; Antisocial Personality Disorder; Recidivism | interventions — Motivational Interviewing; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- brief therapy (Experimental): motivational enhancement therapy for substance use
  Interventions: Behavioral: motivational enhancement therapy
- Standard Care (Placebo Comparator): standard care
  Interventions: Other: standard care

INTERVENTIONS:
Behavioral: motivational enhancement therapy — Four 45-minute MET sessions
  Other Names: SBIRT; brief motivational intervention
  Arms: brief therapy
Other: standard care
  Arms: Standard Care

SUMMARY:
Substance use among criminal offenders constitutes a major public health problem and is tied to negative consequences for offenders, their families, and their communities. One of the direst of these consequences is repeated incarceration; thus, interventions that reduce criminal recidivism are needed. Forensic populations are often viewed with considerable therapeutic pessimism. However, offenders exhibit heterogeneity in personality traits, and the assessment of individual differences among offenders may provide valuable information that guides the use of psychotherapeutic interventions. Among offenders, psychopathy has emerged as an important personality construct for the understanding of violence and criminal recidivism. Moreover, core traits of psychopathy such as lack of empathy, deceitfulness, and lack of remorse may have negative implications for the efficacy of psychosocial interventions. A foundational premise of the present work is that understanding the moderating role of psychopathic traits on substance use treatment outcomes among offenders is essential to determining what works, and for whom. The current proposal is a Phase II randomized clinical trial that aims to examine the impact of psychopathic traits on the efficacy of a brief substance use intervention for offenders in a jail diversion program. Hypotheses that will be examined include: 1) that a Motivational Interviewing (MI) - based treatment will reduce substance use and related consequences relative to a Standard Care only condition, 2) that the reduction in substance use in the intervention group will mediate a reduction in later criminal recidivism relative to the Standard Care condition, and 3) that core psychopathic traits will moderate the efficacy of the intervention such that individuals with lower levels of these traits will derive greater benefits with regard to decreased substance use, decreased drug use consequences, and decreased criminal recidivism at a one-year follow-up.

DETAILED DESCRIPTION:
Substance use among criminal offenders constitutes a major public health problem and is tied to negative consequences for offenders, their families, and their communities. One of the direst of these consequences is repeated incarceration; thus, interventions that reduce criminal recidivism are needed. Forensic populations are often viewed with considerable therapeutic pessimism. However, offenders exhibit heterogeneity in personality traits, and the assessment of individual differences among offenders may provide valuable information that guides the use of psychotherapeutic interventions. Among offenders, psychopathy has emerged as an important personality construct for the understanding of violence and criminal recidivism. Moreover, core traits of psychopathy such as lack of empathy, deceitfulness, and lack of remorse may have negative implications for the efficacy of psychosocial interventions. A foundational premise of the present work is that understanding the moderating role of psychopathic traits on substance use treatment outcomes among offenders is essential to determining what works, and for whom. The current proposal is a Phase II randomized clinical trial that aims to examine the impact of psychopathic traits on the efficacy of a brief substance use intervention for offenders in a jail diversion program. Hypotheses that will be examined include: 1) that a Motivational Interviewing (MI) - based treatment will reduce substance use and related consequences relative to a Standard Care only condition, 2) that the reduction in substance use in the intervention group will mediate a reduction in later criminal recidivism relative to the Standard Care condition, and 3) that core psychopathic traits will moderate the efficacy of the intervention such that individuals with lower levels of these traits will derive greater benefits with regard to decreased substance use, decreased drug use consequences, and decreased criminal recidivism at a one-year follow-up. This work has the potential to provide important data regarding which individuals can benefit from a brief intervention for substance use. Such data will inform the effective and efficient allocation of treatment resources for substance using offenders.

ELIGIBILITY:
Inclusion Criteria:

* In local pretrial services program; English speaking

Exclusion Criteria:

* Psychosis, inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc T. Swogger, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- Pretrial Services, Inc., Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Swogger MT, Conner KR, Caine ED, Trabold N, Parkhurst MN, Prothero LM, Maisto SA. A test of core psychopathic traits as a moderator of the efficacy of a brief motivational intervention for substance-using offenders. J Consult Clin Psychol. 2016 Mar;84(3):248-58. doi: 10.1037/ccp0000065. Epub 2016 Jan 4. PMID 26727409
- See also: PI web page — https://www.urmc.rochester.edu/people/26773384-marc-t-swogger/researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at a jail diversion program in Upstate NY between 2009 and 2014.
Pre-assignment Details: Inclusion criteria were harmful substance use in the past 6 months and enrollment in a jail diversion program subsequent to being charged with a crime.
Groups:
- Standard Care: standard care
  standard care: standard care
Period: Overall Study
Arm/Group | Brief Therapy | Standard Care
Started | 53 | 52
Completed | 39 | 39
Not Completed | 14 | 13
Not completed — Lost to Follow-up | 11 | 11
Not completed — In controlled environment | 3 | 2

BASELINE CHARACTERISTICS:
Population: Participants were adults in an urban pretrial jail diversion program in Upstate New York recruited between 2009 and 2014 subsequent to being charged with a crime.
Groups:
- Brief Motivational Intervention Plus Standard Care (BMI+SC): Brief Motivational Intervention plus Standard Care; Individuals received up to 4 intervention sessions plus assessment and the usual range of services provided by Monroe County Pretrial
- Standard Care (SC): Standard Care: Individuals received assessment only, plus the usual range of services provided by Monroe County Pretrial
- Total: Total of all reporting groups
Arm/Group | Brief Motivational Intervention Plus Standard Care (BMI+SC) | Standard Care (SC) | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (10) | 33.8 (11.8) | 33.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 30 | 38 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 24 | 45
  White | 24 | 26 | 50
  More than one race | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 52 | 105
Psychopathy Checklist-Revised - Factor One (F1) [Mean (Standard Deviation); unit: units on a scale] — The Psychopathy Checklist - Revised is a valid measure of psychopathy with scores ranging from 0-40 (higher indicating higher levels of psychopathy). Factor One of this scale measures interpersonal and affective psychopathic traits and ranges from 0-16.
  units on a scale | 8.1 (4.3) | 9.0 (4.4) | 8.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Days Abstinent Per Month From Drug Use
Description: Using timeline followback data, frequency of substance use was assessed for months three through six and presented as average percent days abstinent per month.
Time Frame: three to six months post baseline
Population: 105 adults (68 men and 37 women) were recruited in an urban pretrial jail diversion program. 78 (74.3%) were retained through six months. Of these, 73 were out of controlled environments (e.g., jail, inpatient treatment) for long enough to have their substance use data analyzed.
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Groups:
- BMI+SC: 1. brief MI + standard care
  2. standard care
- Standard Care: Assessment only plus the usual range of pretrial services
Arm/Group | BMI+SC | Standard Care
Number analyzed (Participants) | 36 | 37
percentage of days abstinent | 46.92 (37.46) | 55.16 (42.09)
Statistical Analysis 1: Comparison: BMI+SC vs Standard Care; A priori hypothesis. Psychopathy Factor 1 (F1) X treatment interaction to predict higher substance use among people high in F1 + who get treatment relative to individuals with high F1 who get standard care; Test type: Superiority or Other; p = .02, Regression, Linear — As stated, the p-value reflects the Factor 1 by treatment interaction term and its effect on percent days abstinent/month

2. Secondary Outcome: Shortened Inventory of Problems With Alcohol and Drugs (SIP-AD)
Description: A measure of consequences of drug and alcohol use across several domains (e.g., social, work, health), SIP-AD scores range from 0-45, with higher scores indicating higher levels of substance use consequences.
Time Frame: six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Therapy | Standard Care
Number analyzed (Participants) | 36 | 37
units on a scale | 10.69 (13.21) | 15.24 (14.28)
Statistical Analysis 1: Comparison: Brief Therapy vs Standard Care; Experimental hypothesis: The F1 X treatment interaction will show that individuals low on F1 who get treatment will reduce substance use consequences at six months relative to those low on F1 who get standard care; Test type: Superiority or Other; p = .34, Regression, Linear — As stated, the p-value reflects the F1 X treatment interaction term and its effect on substance use consequences. A priori threshold for significance was p<.05

3. Secondary Outcome: New Criminal Charge
Description: New criminal charge vs. no new criminal charge at follow-up as indicated by county database.
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | BMI+SC | Standard Care
Number analyzed (Participants) | 36 | 37
participants | 23 | 22
Statistical Analysis 1: Comparison: BMI+SC vs Standard Care; Experimental hypothesis: Treatment X F1 interaction will predict fewer charges at one-year follow-up for individuals low on F1 who got treatment relative to individuals low on F1 who did not; Test type: Superiority or Other; p = .69, Regression, Logistic — a priori threshold p<.05

ADVERSE EVENTS:
Time Frame: Six months from baseline
Description: Criminal recidivism is not considered an adverse event because it is one of the outcome variables. Participants were monitored for serious adverse events through six months of the study (i.e., the last study-related session). There were no adverse events.
Groups:
- Brief Motivational Intervention Plus Standard Care; Standard Care: There were no adverse events for members of this group.
Arm/Group | Brief Motivational Intervention Plus Standard Care | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes